CLINICAL TRIAL: NCT03545802
Title: A Multi-Disciplinary Evaluation of Home-Based High-Intensity Interval Training in People With Type 1 Diabetes: A Pilot Study
Brief Title: Home-HIT and Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Sam Shepherd, Lecturer/Senior Lecturer, Principle Investigator, Liverpool John Moores University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Home-HIT_T1D
Record Dates: First submitted 2018-05-09; First posted 2018-06-04 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training (Experimental): 6 weeks of home-based high intensity interval training
  Interventions: Behavioral: Home-HIT

INTERVENTIONS:
Behavioral: Home-HIT — Participants completed 6 weeks of home-based high-intensity interval training 3 times per week

SUMMARY:
This study aimed to use a multi-disciplinary approach to evaluate a 6-week home-based high-intensity interval training (Home-HIT) intervention in people with type 1 diabetes.

DETAILED DESCRIPTION:
This study aimed to use a multi-disciplinary approach to evaluate a home-based high-intensity interval training (Home-HIT) intervention in people with type 1 diabetes.

Eleven individuals with type 1 diabetes (4 men/7 women; age 30±3 years; BMI 27.1±1.2 kg·m-2; V ̇O2peak 32.4±2.1 ml∙kg∙min-1; duration of type 1 diabetes 10±2 years) completed six weeks of Home-HIT. The effect of Home-HIT on V ̇O2peak, blood pressure, insulin dose and glycaemic profile was assessed pre and post-training. Adherence and ability to meet target heart rate (HR) thresholds (compliance) were monitored using a HR monitor and mobile phone application. Change in glycaemia was measured pre, post and 1h post exercise sessions throughout the six-week period. A qualitative online survey was completed post-training.

This is the first study to combine physiological outcomes with a qualitative evaluation of a training intervention in people with type 1 diabetes. Home-HIT resulted in high adherence alongside increased V ̇O2peak and decreased insulin dose. Because Home-HIT is time-efficient and removes barriers to exercise including fear of hypoglycaemia, it may represent an effective strategy to increase exercise participation in people with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* duration of type 1 diabetes >6 months,
* no significant history of hyper- or hypoglycaemia

Exclusion Criteria:

* duration of type 1 diabetes <6 months,
* significant history of hyper- or hypoglycaemia,
* pregnancy or planning pregnancy,
* uncontrolled hypertension (>180/100 mmHg),
* angina
* autonomic neuropathy,
* taking any medication that affects heart rate (HR)
* major surgery planned within 6 weeks of the study
* severe nonproliferative
* unstable proliferative retinopathy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
change in maximal aerobic capacity | change in baseline maximal aerobic capacity at 6 weeks
  Maximal aerobic capacity was measured pre and post 6 week training intervention using a MOXUS gas analyser on a stationary cycle ergometer
adherence over the course of the training programme | adherence to the training programme over the course of the 6 week intervention
  session completion rate (adherence) was assessed
Compliance over the course of the training programme | compliance to the training programme over the course of the 6 week intervention
  ability to meet target heart rates (compliance) was assessed

SECONDARY OUTCOMES:
change in insulin sensitivity | change in baseline insulin sensitivity at 6 weeks
  insulin dose was recorded pre and post training by participants
change in glycaemic control | change in baseline glycaemic control at 6 weeks
  participants recorded their blood glucose concentrations in the first and final weeks of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
no plan to share

REFERENCES:
- [Derived] Scott SN, Shepherd SO, Andrews RC, Narendran P, Purewal TS, Kinnafick F, Cuthbertson DJ, Atkinson-Goulding S, Noon T, Wagenmakers AJM, Cocks M. A Multidisciplinary Evaluation of a Virtually Supervised Home-Based High-Intensity Interval Training Intervention in People With Type 1 Diabetes. Diabetes Care. 2019 Dec;42(12):2330-2333. doi: 10.2337/dc19-0871. Epub 2019 Sep 17. PMID 31530660